CLINICAL TRIAL: NCT00975650
Title: Efficacy and Tolerability of Nasobol®, an Intra-Nasal Testosterone Product, for Testosterone Replacement in Hypogonadal Men
Brief Title: Efficacy and Tolerability of an Intra-Nasal Testosterone Product
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acerus Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Nasobol-01-2009; TBS1-01
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Hypogonadism
Keywords: Primary Hypogonadism; Secondary Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test 8.0, Ref 5.0, Test 14.0, Test 11.0 (Experimental): Treatment A: 8.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment D: 5.0 mg Androderm® (Positive Control)-Patch, q.d. for 7 days; Treatment C: 14.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment B: 11.0 mg Nasobol® (2 syringes), b.i.d. for 7 days;
  Interventions: Drug: Nasobol®; Drug: Androderm® (Positive Control)
- Test 11.0, Test 8.0, Ref 5.0, Test 14.0 (Experimental): Treatment B: 11.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment A: 8.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment D: 5.0 mg Androderm® (Positive Control)-Patch, q.d. for 7 days; Treatment C: 14.0 mg Nasobol® (2 syringes), b.i.d. for 7 days
  Interventions: Drug: Nasobol®; Drug: Androderm® (Positive Control)
- Test 14.0, Test 11.0, Test 8.0, Ref 5.0 (Experimental): Treatment C: 14.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment B: 11.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment A: 8.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment D: 5.0 mg Androderm® (Positive Control)-Patch, q.d. for 7 days;
  Interventions: Drug: Nasobol®; Drug: Androderm® (Positive Control)
- Ref 5.0, Test 14.0, Test 11.0, Test 8.0 (Experimental): Treatment D: 5.0 mg Androderm® (Positive Control)-Patch, q.d. for 7 days; Treatment C: 14.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment B: 11.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment A: 8.0 mg Nasobol® (2 syringes), b.i.d. for 7 days
  Interventions: Drug: Nasobol®; Drug: Androderm® (Positive Control)

INTERVENTIONS:
Drug: Nasobol® — Intra-nasal Testosterone (2 syringes), b.i.d.
Drug: Androderm® (Positive Control) — QD administration

SUMMARY:
This clinical trial is being performed to compare the pharmacokinetic profile of testosterone after repeated intra-nasal administration of products of different strengths in subjects with hypogonadism.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective of this study was to determine the efficacy of Nasobol in the treatment of hypogonadal men requiring testosterone replacement therapy. Efficacy was determined by establishing a pharmacokinetic profile for serum testosterone levels following Nasobol treatment, and comparing it to that of the active control, Androderm®.

Secondary Objective:

To establish a safety profile for Nasobol.

ELIGIBILITY:
Inclusion Criteria:

* Men with primary or secondary hypogonadism and a serum morning (0900 h ± 30 minutes) testosterone levels >100 ng/dl and ≤ 300 ng/dL.
* Normal Otolaryngological nasal endoscopy examination.
* Normal prostate examination (no palpable prostatic mass), and serum PSA ≤ 4.0 ng/mL.

Exclusion Criteria:

* Current treatment with other androgens (i.e. DHEA), anabolic steroids or other sex hormones
* Treatment with Estrogens, GnRH antagonists, or Growth Hormone within previous 12 months
* History of nasal surgery, specifically turbinoplasty, septoplasty, rhinoplasty, or sinus surgery.
* History of nasal disorders (e.g. polyposis, recurrent epistaxis ( > 1 nose bleed per month, abuse of nasal decongestants) or sleep apnea.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Desjardins, Ph.D, Study Director — Trimel Biopharma
Locations (6):
- United States (6):
  - Quality of Life Medical & Research centre, Tucson, Arizona
  - Providence Clinical Research, Burbank, California
  - Cetero Research, Miami Gardens, Florida
  - Clinical Research Institute, Wichita, Kansas
  - Regional Urology, LLC, Shreveport, Louisiana
  - dgd Research Inc., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Treatment A: 8.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment D: 5.0 mg Androderm® (Positive Control)-Patch, q.d. for 7 days; Treatment C: 14.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment B: 11.0 mg Nasobol® (2 syringes), b.i.d. for 7 days;
- Sequence 2: Treatment B: 11.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment A: 8.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment D: 5.0 mg Androderm® (Positive Control)-Patch, q.d. for 7 days; Treatment C: 14.0 mg Nasobol® (2 syringes), b.i.d. for 7 days
- Sequence 3: Treatment C: 14.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment B: 11.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment A: 8.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment D: 5.0 mg Androderm® (Positive Control)-Patch, q.d. for 7 days
- Sequence 4: Treatment D: 5.0 mg Androderm® (Positive Control)-Patch, q.d. for 7 days; Treatment C: 14.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment B: 11.0 mg Nasobol® (2 syringes), b.i.d. for 7 days; Treatment A: 8.0 mg Nasobol® (2 syringes), b.i.d. for 7 days
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 13 | 16 | 14 | 14
Completed | 13 | 16 | 14 | 14
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 13 | 16 | 14 | 14
Completed | 12 | 14 | 14 | 14
Not Completed | 1 | 2 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 12 | 14 | 14 | 14
Completed | 12 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 12 | 14 | 14 | 14
Completed | 12 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All Subjects who were dosed.
Arm/Group | All Subjects
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 53
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Serum Testosterone Ln-Cmax
Description: The primary objective of this study was to determine the efficacy of Nasobol in the treatment of hypogonadal men requiring testosterone replacement therapy. Efficacy was determined by establishing a pharmacokinetic profile for serum testosterone levels following Nasobol treatment or that of the active control, Androderm®.
Time Frame: 0.0 (trough), 0.50, 1.0, 1.5, 2.0, 3.0, 6.0, 9.0, 10.0, 10.5, 11.0, 11.5, 12.0, 13.0, 16.0, 19.0, 22.0, and 24.0 hours.
Population: Number of participants includes participants who completed the corresponding treatment and had sufficient plasma concentration data to calculate the PK parameter.
Measure: Mean (Standard Deviation); unit: ng/dL
Groups:
- Treatment A: Treatment A: 8.0 mg Nasobol® (2 syringes), b.i.d. for 7 days
- Treatment B: Treatment B: 11.0 mg Nasobol® (2 syringes), b.i.d. for 7 days
- Treatment C: Treatment C: 14.0 mg Nasobol® (2 syringes), b.i.d. for 7 days
- Treatment D: Treatment D: 5.0 mg Androderm® (Positive Control)-Patch, q.d. for 7 days
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 52 | 55 | 52 | 54
ng/dL | 6.25 (0.37) | 6.41 (0.35) | 6.54 (0.36) | 6.36 (0.37)

2. Primary Outcome: Serum Testosterone Ln-AUCt
Time Frame: 0.0 (trough), 0.50, 1.0, 1.5, 2.0, 3.0, 6.0, 9.0, 10.0, 10.5, 11.0, 11.5, 12.0, 13.0, 16.0, 19.0, 22.0, and 24.0 hours.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/dL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 52 | 55 | 52 | 54
ng.h/dL | 8.80 (0.26) | 8.90 (0.27) | 8.95 (0.29) | 9.09 (0.29)

3. Primary Outcome: Serum Testosterone Cavg
Time Frame: 0.0 (trough), 0.50, 1.0, 1.5, 2.0, 3.0, 6.0, 9.0, 10.0, 10.5, 11.0, 11.5, 12.0, 13.0, 16.0, 19.0, 22.0, and 24.0 hours.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 52 | 55 | 52 | 54
ng/dL | 287.10 (76.42) | 316.64 (88.93) | 336.11 (100.76) | 384.62 (102.97)

4. Primary Outcome: Serum Dihydrotestosterone Ln-Cmax
Time Frame: 0.0 (trough), 0.50, 1.0, 1.5, 2.0, 3.0, 6.0, 9.0, 10.0, 10.5, 11.0, 11.5, 12.0, 13.0, 16.0, 19.0, 22.0, and 24.0 hours.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 52 | 55 | 52 | 54
ng/dL | 3.54 (0.38) | 3.67 (0.44) | 3.80 (0.41) | 3.44 (0.35)

5. Primary Outcome: Serum Dihydrotestosterone Ln-AUCt
Time Frame: 0.0 (trough), 0.50, 1.0, 1.5, 2.0, 3.0, 6.0, 9.0, 10.0, 10.5, 11.0, 11.5, 12.0, 13.0, 16.0, 19.0, 22.0, and 24.0 hours.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/dL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 52 | 55 | 52 | 54
ng.h/dL | 6.34 (0.38) | 6.47 (0.41) | 6.52 (0.45) | 6.33 (0.34)

6. Primary Outcome: Serum Dihydrotestosterone Cavg
Time Frame: 0.0 (trough), 0.50, 1.0, 1.5, 2.0, 3.0, 6.0, 9.0, 10.0, 10.5, 11.0, 11.5, 12.0, 13.0, 16.0, 19.0, 22.0, and 24.0 hours.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 52 | 55 | 52 | 54
ng/dL | 25.24 (8.51) | 28.97 (11.41) | 30.79 (12.50) | 24.69 (8.46)

7. Primary Outcome: Percentage of Subjects With Cavg Within the Reference Range
Description: The percentage of subjects with a Cavg within the reference range of 300 to 1050 ng/dL and 25.5 to 97.8 ng/dL for testosterone and dihydotestosterone.
Time Frame: Each period is 7 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 52 | 55 | 52 | 54
Participants
  Testosterone | 19 | 27 | 27 | 42
  Dihydrotestosterone | 24 | 31 | 34 | 22

ADVERSE EVENTS:
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/56 | 0/54 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56 | 0/54 | 0/55
Other Adverse Events (participants affected / at risk) | 5/57 | 6/56 | 0/54 | 6/55
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=57) | Treatment B (N=56) | Treatment C (N=54) | Treatment D (N=55)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Application Site Rash (General disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 2 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No